CLINICAL TRIAL: NCT05649059
Title: Investigating the Effects of Cannabidiol on Social Anxiety Disorder
Acronym: CAN-SAD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts Institute of Technology (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2206000688
Record Dates: First submitted 2022-11-30; First posted 2022-12-13 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Phobia, Social
Keywords: Social Anxiety Disorder; Cannabidiol; fMRI
MeSH Terms: conditions — Phobia, Social | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (Active Comparator): 300mg Cannabidiol (3mL Epidiolex), oral, single-dose
  Interventions: Drug: Cannabidiol
- Placebo (Placebo Comparator): Placebo (3mL sesame seed oil), oral, single-dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol — Participants randomized to the cannabidiol arm will receive 3mL of Epidiolex (100mg cannabidiol/mL) in a single-dose.
  Other Names: Epidiolex
  Arms: Cannabidiol
Drug: Placebo — Participants randomized to the placebo arm will receive 3mL of placebo (sesame seed oil) in a single dose.
  Arms: Placebo

SUMMARY:
The purpose of this study is to test whether a single-dose of Epidiolex (cannabidiol) is associated with reduced psychological, physiological, and neuroimaging measures of anxiety in people diagnosed with social anxiety disorder (SAD).

DETAILED DESCRIPTION:
Using a randomized, double-blind, placebo-controlled, parallel-group study design, this scientific investigation will examine the effect of 3 milliliters (mL) of Epidiolex (100mg cannabidiol/mL) on behavioral, physiological, and neuroimaging measures of anxiety in subjects diagnosed with SAD. The study will enroll 50 subjects with SAD who will be randomized in a double-blind manner to receive either Epidiolex or placebo before experiencing the Trier Social Stress Test (TSST), the gold-standard for ethically inducing stress in a controlled laboratory setting. Following the TSST, neuroimaging measures of emotional processing and self-referential processing will be acquired using functional magnetic resonance imaging (fMRI).

This study will be conducted primarily at Massachusetts Institute of Technology with research and clinical support from Massachusetts General Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to provide written informed consent.
* Sufficiently fluent in English to participate in the trial.
* Between 18-55 years of age (inclusive).
* Right-hand dominant.
* Current medications are stable for past 30 days (no changes to dose or frequency).
* Negative result on pregnancy test (if female).
* Negative result on urine drug screening.
* Liebowitz Social Anxiety Scale (LSAS ≥ 60).

Exclusion Criteria:

* History of bipolar disorder, schizophrenia, psychosis, delusional disorders.
* History of eating disorder within past 6 months.
* History of any traumatic brain injury.
* Currently diagnosed with diabetes mellitus.
* Presence of severe medical illness that would prevent completion of study procedures.
* Presence of significant neurological illness or cognitive dysfunction (e.g.; seizures, dementia).
* History of substance use disorder within past 6 months (other than nicotine and caffeine).
* Use of any cannabis-containing products in past 30 days (CBD or THC).
* Use of benzodiazepines in past 2 weeks.
* Use of alpha- or beta-blockers in past week.
* History of claustrophobia.
* Contraindications for MRI (e.g.; shrapnel).
* Presence of any other medical condition that, in the investigator's opinion, may interfere with the study procedures.
* Use of concomitant medication that has a strong interaction with CBD.
* History of liver disease.
* History of hypersensitivity to cannabinoids.
* History of hypersensitivity to sesame seed oil.
* Currently breastfeeding (if female).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in Acute Subjective Anxiety | -180 minutes, -15 minutes, -5 minutes, +10 minutes, +20 minutes, +30 minutes
  Subjective anxiety will be assessed with a modified Visual Analog Mood Scale (VAMS) which utilizes a vertical 100 millimeter (mm) bipolar visual scale between two opposing moods consisting of the following word pairs: calm-excited, relaxed-tense, and tranquil-troubled. Total subjective anxiety for each timepoint will be the average distance from the top for the three-question battery. VAMS will be assessed 15 minutes before drug administration (-180 minutes before start of TSST), 150 minutes after drug administration (-15 minutes before start of TSST), after the Anticipation Phase (-5 minutes before start of TSST), after the Stress Procedures (+10 minutes after start of TSST), after 5 minutes in the Recovery Phase (+20 minutes after start of TSST), and 15 minutes after start of the Recovery Phase (+30 minutes after start of TSST).

SECONDARY OUTCOMES:
Differences in Salivary Alpha Amylase | -180 minutes, -15 minutes, -5 minutes, +10 minutes, +20 minutes, +30 minutes
  Physiological stress will be assessed indirectly with salivary alpha amylase (sAA) activity which is regulated by the sympathetic branch of the autonomic nervous system. Samples will be collected using the SalivaBio Oral Swab (SOS) from Salimetrics. Participants will place the SOS in their mouth for 1-2 minutes at each timepoint to collect saliva. sAA will be assessed 15 minutes before drug administration (-180 minutes before start of TSST), 150 minutes after drug administration (-15 minutes before start of TSST), after the Anticipation Phase (-5 minutes before start of TSST), after the Stress Procedures (+10 minutes after start of TSST), after 5 minutes in the Recovery Phase (+20 minutes after start of TSST), and 15 minutes after start of the Recovery Phase (+30 minutes after start of TSST).

OTHER OUTCOMES:
Differences in fMRI BOLD Response | +45 minutes
  Patterns of brain activation measured as blood-oxygenation-level dependent (BOLD) signals will be assessed using 3.0 Tesla (3T) functional magnetic resonance imaging (fMRI). Several exploratory imaging paradigms, including the emotional face-matching task (EFMT) and the self-referential comment task (SRCT), will be used to examine differences between participants who receive Epidiolex (cannabidiol) and those that receive placebo. Neuroimaging will begin approximately 210 minutes after drug administration (+45 minutes after the TSST).

CONTACTS AND LOCATIONS:
Overall Officials: John Gabrieli, PhD, Principal Investigator — Massachusetts Institute of Technology
Locations (1):
- Massachusetts Institute of Technology, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
All data, code, and materials used in the analyses will be made available upon request by John Gabrieli and Massachusetts Institute of Technology after scientific review and a completed data use agreement/material transfer agreement beginning one year after publication of the results. Any requests should be submitted to John Gabrieli at gabrieli@mit.edu.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will become available beginning one year after publication of the results.
Access Criteria: Data will be provided pending a scientific review and a completed data use agreement/material transfer agreement. Requests should be submitted to John Gabrieli at gabrieli@mit.edu.

REFERENCES:
- See also: CAN-SAD Recruitment Site — https://redcap.link/CANSAD